CLINICAL TRIAL: NCT00679588
Title: A Multinational, Multicenter, Randomized, Double Blind Study Comparing the Efficacy and Safety of AVE5026 With Enoxaparin for the Prevention of Venous Thromboembolism in Patients Undergoing Major Abdominal Surgery
Brief Title: Evaluation of AVE5026 as Compared to Enoxaparin for the Prevention of Venous Thromboembolism in Patients Undergoing Major Abdominal Surgery
Acronym: SAVE-ABDO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC6520; 2007-007942-36 (EudraCT Number)
Record Dates: First submitted 2008-05-07; First posted 2008-05-19 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-11

CONDITIONS: Venous Thromboembolism
Keywords: Digestive System Surgical Procedure; Urologic Surgical Procedure; Prevention of venous thromboembolism; Abdominal surgery
MeSH Terms: conditions — Venous Thromboembolism | interventions — AVE 5026; enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semuloparin (Experimental): Semuloparin sodium 20 mg (10 mg if Severe Renal Impairment [SRI]) once daily for 7-10 days with an initial dose given 8 hours after surgery (placebo for Enoxaparin sodium prior to surgery according to local standard for Enoxaparin and 12 hours after surgery to maintain the blind)
  Interventions: Drug: Semuloparin Sodium; Drug: Placebo
- Enoxaparin (Active Comparator): Enoxaparin sodium 40 mg (20 mg if Severe Renal Impairment [SRI]) once daily for 7-10 days with an initial dose given prior to or 12 hours after surgery according to local standard for Enoxaparin sodium (placebo for Semuloparin sodium 8 hours after surgery to maintain the blind)
  Interventions: Drug: Enoxaparin sodium; Drug: Placebo

INTERVENTIONS:
Drug: Semuloparin Sodium — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection
  Other Names: AVE5026
  Arms: Semuloparin
Drug: Enoxaparin sodium — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection
  Other Names: Lovenox®
  Arms: Enoxaparin
Drug: Placebo — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml prefilled syringe strictly identical in appearance containing the same volume but without active component
  Subcutaneous injection

SUMMARY:
The primary objective is to compare the efficacy and safety of once daily (q.d.) subcutaneous (s.c.) injections of Semuloparin sodium (AVE5026) with q.d. s.c. injections of Enoxaparin for the prevention of Venous Thromboembolic Events (VTE) in patients undergoing major abdominal surgery.

The secondary objectives are to evaluate the safety of Semuloparin sodium (AVE5026) and to document Semuloparin sodium (AVE5026) exposure in this population.

DETAILED DESCRIPTION:
Randomization has to take place prior to the surgery.

The total duration of observation per participant is 35-42 days from surgery broken down as follows:

* 7 to 10-day double-blind treatment period;
* 28 to 35-day follow-up period.

Mandatory bilateral venography of the lower limbs has to be performed between 7 to 11 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing major abdominal surgery (open surgery under general anesthesia lasting more than 45 minutes in the peritoneal and/or retroperitoneal space and/or pelvis).
* Patient <60 years of age had to have one of the following additional risk factors for VTE:

  * History of VTE,
  * Obesity,
  * Chronic Heart failure,
  * Chronic Respiratory Failure,
  * Inflammatory Bowel Disease,
  * Cancer Surgery.

Exclusion Criteria:

* Any major orthopedic or general surgery in the 3 months prior to study start;
* Clinical signs or symptoms of DVT or PE within the last 12 months or known post phlebitic syndrome;
* Any contra-indications to the performance of venography;
* High risk of bleeding;
* Known hypersensitivity to heparin or Enoxaparin sodium;
* End stage renal disease or patient on dialysis.

The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4413 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experience Venous Thromboembolism Event (VTE) or All-cause Death | From randomization up to 10 days after surgery or the day of mandatory venography, whichever comes first
  VTE includes any proximal or distal Deep Vein Thrombosis (DVT) (symptomatic or not) and non-fatal Pulmonary Embolism (PE) as confirmed by a Central Independent Adjudication Committee (CIAC) after review of mandatory bilateral venograms and diagnostic tests for VTE.
  All-cause deaths includes fatal PE and deaths for other reason than PE.

SECONDARY OUTCOMES:
Percentage of Participants Who Experience "major" VTE or All-cause Death | From randomization up to 10 days after surgery or the day of mandatory venography, whichever comes first
  "major" VTE includes any proximal DVT, symptomatic distal DVT and non-fatal Pulmonary Embolism (PE) as as confirmed by the CIAC.
Percentage of Participants Who Experience Clinically Relevant Bleedings ("major" and "clinically relevant non-major" bleedings ) | From 1st study drug injection up to 3 days after last study drug injection
  Bleedings are centrally and blindly reviewed by the CIAC and classified as:
  * "major" (fatal, in a critical area/organ, causing a post-operative drop in hemoglobin ≥2 g/dL or requiring post-operative transfusion ≥2 units of blood, leading to an invasive diagnostic or therapeutic intervention, or associated with circulatory decompensation);
  * "clinically relevant non-major" (skin hematoma or epistaxis requiring surgical/medical intervention/treatment, macroscopic hematuria, or overt bleeding requiring specific attention by health care professional);
  * "Nonclinically relevant bleeding".
Percentage of Participants requiring the initiation of curative anticoagulant or thrombolytic treatment after VTE assessment | From randomization up to 10 days after surgery or the day of mandatory venography, whichever comes first
  Initiation of curative anticoagulant or thrombolytic treatment after VTE assessment was defined from investigator's answer to the question "was the subject treated for VTE?" asked after the diagnostic tests for suspected VTE and after the mandatory venography.

OTHER OUTCOMES:
Number of Deaths on Treatment | From 1st study drug injection up to 3 days after last study drug injection
  All deaths are centrally and blindly reviewed by the CIAC and classified as fatal PE, fatal bleeding, cardiovascular death or other based on relevant documentation (e.g. autopsy report).
Platelets Count: Percentage of Participants With Potentially Clinically Significant Abnormalities (PCSA) | From 1st study drug injection up to 3 days after last study drug injection
  PCSA are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review.
  Thresholds for platelet counts are defined as <100 Giga/L.
Liver Function: Percentage of Participants With Potentially Clinically Significant Abnormalities (PCSA) | From 1st study drug injection up to 3 days after last study drug injection
  Thresholds are defined as follows:
  * Alanine Aminotransferase (ALT) >3 Upper Normal Limit (ULN);
  * Total Bilirubin (TB) >2 ULN;
  * ALT >3 ULN and TB >2 ULN;
  Cases with ALT >3 ULN and TB >2 ULN (not necessarily concomitant) are evaluated by a blinded independent adjudicator to determine if they met Hy's law criteria.
Trough Plasma Concentration of Semuloparin Sodium (AVE5026) | 0.5-1 and 2-4 hours after Day 1 first post-operative injection, 6-8 and 10-16 hours after Day 4 injection, and just before the last injection
  Trough Plasma Concentration [Ctrough] is defined as plasma concentrations obtained just before study drug injection (i.e.24h±2h after study drug injection).
  Lower Limit Of Quantification (LLOQ) is defined as 0,348 μgEq/mL. Concentrations below LLOQ are replaced by half of LLOQ for the calculation.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kakkar, Prof., MD, PhD, Principal Investigator — Queen Mary's School of Medicine & Dentistry, London (UK); Alexander Turpie, MD, Study Chair — HHS-General Hospital, Hamilton, Canada
Locations (270):
- United States (25):
  - Investigational Site Number 840026, Birmingham, Alabama
  - Investigational Site Number 840035, Birmingham, Alabama
  - Investigational Site Number 840042, Birmingham, Alabama
  - Investigational Site Number 840002, Birmingham, Alabama
  - Investigational Site Number 840031, Corlton, California
  - Investigational Site Number 840007, Huntingdon Beach, California
  - Investigational Site Number 840014, Los Angeles, California
  - Investigational Site Number 840011, Sant Barbara, California
  - Investigational Site Number 840021, Denver, Colorado
  - Investigational Site Number 840029, Clearwater, Florida
  - Investigational Site Number 840017, Jacksonville, Florida
  - Investigational Site Number 840044, Miami, Florida
  - Investigational Site Number 840015, Orlando, Florida
  - Investigational Site Number 840009, Columbus, Georgia
  - Investigational Site Number 840019, Maywood, Illinois
  - Investigational Site Number 840036, Springfield, Illinois
  - Investigational Site Number 840037, Hazard, Kentucky
  - Investigational Site Number 840008, St Louis, Missouri
  - Investigational Site Number 840020, Teaneck, New Jersey
  - Investigational Site Number 840051, Columbus, Ohio
  - Investigational Site Number 840006, Pittsburgh, Pennsylvania
  - Investigational Site Number 840025, Houston, Texas
  - Investigational Site Number 840050, Houston, Texas
  - Investigational Site Number 840032, Lubbock, Texas
  - Investigational Site Number 840043, Morgantown, West Virginia
- Argentina (8):
  - Investigational Site Number 032002, Buenos Aires
  - Investigational Site Number 032001, Buenos Aires
  - Investigational Site Number 032004, Buenos Aires
  - Investigational Site Number 032007, Capital Federal
  - Investigational Site Number 032008, Capital Federal
  - Investigational Site Number 032014, Córdoba
  - Investigational Site Number 032012, Rosario
  - Investigational Site Number 032005, Santa Fe
- Australia (4):
  - Investigational Site Number 036002, Box Hill
  - Investigational Site Number 036003, Box Hill
  - Investigational Site Number 036001, Kogarah
  - Investigational Site Number 036008, Redcliffe
- Austria (2):
  - Investigational Site Number 040001, Graz
  - Investigational Site Number 040002, Wels
- Belarus (8):
  - Investigational Site Number 112001, Homyel
  - Investigational Site Number 112006, Homyel
  - Investigational Site Number 112003, Minsk
  - Investigational Site Number 112008, Minsk
  - Investigational Site Number 112002, Minsk
  - Investigational Site Number 112005, Minsk
  - Investigational Site Number 112004, Vitebsk
  - Investigational Site Number 112007, Vitebsk
- Belgium (2):
  - Investigational Site Number 056002, Genk
  - Investigational Site Number 056001, Ghent
- Brazil (14):
  - Investigational Site Number 076003, Belo Horizonte
  - Investigational Site Number 076010, Belo Horizonte
  - Investigational Site Number 076014, Caxias do Sul
  - Investigational Site Number 076012, Curitiba
  - Investigational Site Number 076005, Curitiba
  - Investigational Site Number 076006, Goiânia
  - Investigational Site Number 076011, Joinville
  - Investigational Site Number 076007, Porto Alegre
  - Investigational Site Number 076009, Porto Alegre
  - Investigational Site Number 076015, Ribeirão Preto
  - Investigational Site Number 076013, São José do Rio Preto
  - Investigational Site Number 076004, São Paulo
  - Investigational Site Number 076002, São Paulo
  - Investigational Site Number 076008, São Paulo
- Bulgaria (8):
  - Investigational Site Number 100004, Pleven
  - Investigational Site Number 100003, Rousse
  - Investigational Site Number 100011, Sofia
  - Investigational Site Number 100005, Sofia
  - Investigational Site Number 100008, Sofia
  - Investigational Site Number 100009, Sofia
  - Investigational Site Number 100006, Varna
  - Investigational Site Number 100010, Varna
- Canada (7):
  - Investigational Site Number 124001, Edmonton
  - Investigational Site Number 124004, Kitchener
  - Investigational Site Number 124010, Montreal
  - Investigational Site Number 124011, Red Deer
  - Investigational Site Number 124009, Saint John
  - Investigational Site Number 124002, Thunder Bay
  - Investigational Site Number 124007, Vancouver
- Chile (2):
  - Investigational Site Number 152002, Rancagua
  - Investigational Site Number 152001, Santiago
- China (11):
  - Investigational Site Number 156011, Baotou
  - Investigational Site Number 156012, Changsha
  - Investigational Site Number 156010, Changsha
  - Investigational Site Number 156006, Fuzhou
  - Investigational Site Number 156003, Guangzhou
  - Investigational Site Number 156013, Haikou
  - Investigational Site Number 156005, Nanjing
  - Investigational Site Number 156008, Qingdao
  - Investigational Site Number 156001, Shijiazhuang
  - Investigational Site Number 156014, Tianjin
  - Investigational Site Number 156004, Xi'an
- Croatia (3):
  - Investigational Site Number 191004, Požega
  - Investigational Site Number 191001, Pula
  - Investigational Site Number 191002, Zagreb
- Czechia (14):
  - Investigational Site Number 203007, Brno
  - Investigational Site Number 203001, Brno
  - Investigational Site Number 203011, Jihlava
  - Investigational Site Number 203015, Kolín
  - Investigational Site Number 203009, Kroměříž
  - Investigational Site Number 203004, Liberec
  - Investigational Site Number 203014, Most
  - Investigational Site Number 203003, Ostrava
  - Investigational Site Number 203012, Pardubice
  - Investigational Site Number 203008, Prague
  - Investigational Site Number 203006, Prague
  - Investigational Site Number 203002, Prague
  - Investigational Site Number 203016, Říčany
  - Investigational Site Number 203010, Ústí nad Labem
- Denmark (2):
  - Investigational Site Number 208001, København NV
  - Investigational Site Number 208002, Odense C
- Estonia (3):
  - Investigational Site Number 233003, Tallinn
  - Investigational Site Number 233001, Tartu
  - Investigational Site Number 233002, Tartu
- Germany (11):
  - Investigational Site Number 276011, Bochum
  - Investigational Site Number 276015, Castrop-Rauxel
  - Investigational Site Number 276018, Castrop-Rauxel
  - Investigational Site Number 276006, Dresden
  - Investigational Site Number 276012, Hanover
  - Investigational Site Number 276002, Heidelberg
  - Investigational Site Number 276004, Homburg
  - Investigational Site Number 276014, Lübeck
  - Investigational Site Number 276016, Magdeburg
  - Investigational Site Number 276013, München
  - Investigational Site Number 276001, Stralsund
- Investigational Site Number 300002, Heraklion, Greece
- Hungary (5):
  - Investigational Site Number 348007, Debrecen
  - Investigational Site Number 348009, Kistarcsa
  - Investigational Site Number 348008, Szeged
  - Investigational Site Number 348004, Székesfehérvár
  - Investigational Site Number 348003, Szolnok
- India (29):
  - Investigational Site Number 356005, Ahmedabad
  - Investigational Site Number 356004, Ahmedabad
  - Investigational Site Number 356033, Andhra Pradesh
  - Investigational Site Number 356011, Bangalore
  - Investigational Site Number 356027, Bangalore
  - Investigational Site Number 356008, Bangalore
  - Investigational Site Number 356019, Banglore
  - Investigational Site Number 356031, Bhopal
  - Investigational Site Number 356014, Chennai
  - Investigational Site Number 356018, Chennai
  - Investigational Site Number 356016, Chennai
  - Investigational Site Number 356021, Chennai
  - Investigational Site Number 356006, Coimbatore
  - Investigational Site Number 356025, Gujarat
  - Investigational Site Number 356028, Hyderabad
  - Investigational Site Number 356010, Hyderabad
  - Investigational Site Number 356002, Jaipur
  - Investigational Site Number 356022, Jaipur
  - Investigational Site Number 356013, Kochi
  - Investigational Site Number 356007, Kochi
  - Investigational Site Number 356003, Lucknow
  - Investigational Site Number 356026, Lucknow
  - Investigational Site Number 356032, Ludhiana
  - Investigational Site Number 356001, Mangalore
  - Investigational Site Number 356030, Nagpur
  - Investigational Site Number 356009, New Delhi
  - Investigational Site Number 356023, Pune
  - Investigational Site Number 356015, Pune
  - Investigational Site Number 356012, Punjgutta
- Italy (11):
  - Investigational Site Number 380009, Aviano
  - Investigational Site Number 380001, Genova
  - Investigational Site Number 380015, Genova
  - Investigational Site Number 380006, Milan
  - Investigational Site Number 380004, Padua
  - Investigational Site Number 380008, Parma
  - Investigational Site Number 380013, Piacenza
  - Investigational Site Number 380012, Pordenone
  - Investigational Site Number 380005, Reggio Emilia
  - Investigational Site Number 380011, San Donato Milanese
  - Investigational Site Number 380007, Trieste
- Latvia (3):
  - Investigational Site Number 428004, Daugavpils
  - Investigational Site Number 428003, Riga
  - Investigational Site Number 428002, Riga
- Lithuania (3):
  - Investigational Site Number 440003, Kaunas
  - Investigational Site Number 440001, Kaunas
  - Investigational Site Number 440002, Vilnius
- Mexico (2):
  - Investigational Site Number 484001, Guadalajara
  - Investigational Site Number 484006, Mazatlán
- New Zealand (3):
  - Investigational Site Number 554003, Christchurch
  - Investigational Site Number 554001, Christchurch
  - Investigational Site Number 554002, Nelson South
- Investigational Site Number 578001, Trondheim, Norway
- Peru (6):
  - Investigational Site Number 604003, Callao
  - Investigational Site Number 604004, Callao
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604001, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604002, Lima
- Poland (18):
  - Investigational Site Number 616001, Bydgoszcz
  - Investigational Site Number 616003, Bydgoszcz
  - Investigational Site Number 616006, Gdansk
  - Investigational Site Number 616005, Krakow
  - Investigational Site Number 616018, Krakow
  - Investigational Site Number 616020, Krakow
  - Investigational Site Number 616009, Lodz
  - Investigational Site Number 616002, Lodz
  - Investigational Site Number 616010, Lublin
  - Investigational Site Number 616012, Poznan
  - Investigational Site Number 616015, Sosnowiec
  - Investigational Site Number 616013, Szczecin
  - Investigational Site Number 616011, Torun
  - Investigational Site Number 616004, Warsaw
  - Investigational Site Number 616014, Warsaw
  - Investigational Site Number 616008, Wroclaw
  - Investigational Site Number 616007, Wroclaw
  - Investigational Site Number 616016, Wroclaw
- Romania (6):
  - Investigational Site Number 642003, Cluj-Napoca
  - Investigational Site Number 642006, Cluj-Napoca
  - Investigational Site Number 642005, Cluj-Napoca
  - Investigational Site Number 642001, Oradea
  - Investigational Site Number 642004, Oradea
  - Investigational Site Number 642002, Timișoara
- Russia (20):
  - Investigational Site Number 643019, Krasnodar
  - Investigational Site Number 643006, Krasnoyarsk
  - Investigational Site Number 643003, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643020, Moscow
  - Investigational Site Number 643021, Moscow
  - Investigational Site Number 643025, Moscow
  - Investigational Site Number 643008, Novosibirsk
  - Investigational Site Number 643007, Novosibirsk
  - Investigational Site Number 643026, Omsk
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643010, Saint Petersburg
  - Investigational Site Number 643009, Saint Petersburg
  - Investigational Site Number 643018, Saint Petersburg
  - Investigational Site Number 643017, Saint Petersburg
  - Investigational Site Number 643015, Sestroretsk
  - Investigational Site Number 643012, Tomsk
  - Investigational Site Number 643016, Vsevolozhsk
  - Investigational Site Number 643014, Yaroslavl
- Serbia (3):
  - Investigational Site Number 688001, Belgrade
  - Investigational Site Number 688004, Belgrade
  - Investigational Site Number 688002, Novi Sad
- Investigational Site Number 703001, Bratislava, Slovakia
- Slovenia (2):
  - Investigational Site Number 705001, Celje
  - Investigational Site Number 705002, Maribor
- South Africa (3):
  - Investigational Site Number 710001, Cape Town
  - Investigational Site Number 710004, Cape Town
  - Investigational Site Number 710003, Worcester
- South Korea (10):
  - Investigational Site Number 410007, Daegu
  - Investigational Site Number 410006, Goyang
  - Investigational Site Number 410001, Gyeonggi-do
  - Investigational Site Number 410009, Incheon
  - Investigational Site Number 410011, Seoul
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410010, Seoul
  - Investigational Site Number 410008, Seoul
  - Investigational Site Number 410003, Suwon
- Spain (2):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724002, Madrid
- Sweden (4):
  - Investigational Site Number 752002, Kungälv
  - Investigational Site Number 752004, Norrköping
  - Investigational Site Number 752001, Stockholm
  - Investigational Site Number 752003, Varberg
- Turkey (Türkiye) (4):
  - Investigational Site Number 792003, Istanbul
  - Investigational Site Number 792001, Istanbul
  - Investigational Site Number 792006, Istanbul
  - Investigational Site Number 792007, Izmir
- Ukraine (8):
  - Investigational Site Number 804003, Cherkasy
  - Investigational Site Number 804007, Donetsk
  - Investigational Site Number 804010, Donetsk
  - Investigational Site Number 804011, Kharkiv
  - Investigational Site Number 804005, Kyiv
  - Investigational Site Number 804002, Kyiv
  - Investigational Site Number 804004, Kyiv
  - Investigational Site Number 804008, Odesa
- Investigational Site Number 826001, London, United Kingdom

REFERENCES:
- [Derived] Kakkar AK, Agnelli G, Fisher W, George D, Lassen MR, Mismetti P, Mouret P, Murphy J, Lawson F, Turpie AG; SAVE-ABDO Investigators. Preoperative enoxaparin versus postoperative semuloparin thromboprophylaxis in major abdominal surgery: a randomized controlled trial. Ann Surg. 2014 Jun;259(6):1073-9. doi: 10.1097/SLA.0000000000000430. PMID 24374549